CLINICAL TRIAL: NCT06920602
Title: Development and Evaluation of an AI-empowered Voice-interactive Chatbot for Migraine Management Among Hong Kong Women: a Randomized Crossover Trial
Brief Title: AI Chatbot for Migraine Management in Hong Kong Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Nethersole Institute of Continuing Holistic Health Education (NICHE) (Unknown)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HSEARS20241015007; RG2024/2025_A_11 (Other Grant/Funding Number: NICHE)
Record Dates: First submitted 2025-03-10; First posted 2025-04-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-04

CONDITIONS: Migraine
Keywords: migraine; RCT; migraine diary; artificial intelligence; chatbot
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): AI-empowered voice-interactive chatbot followed by paper migraine diary
  Interventions: Device: AI-empowered voice-interactive chatbot; Device: Paper migraine diary
- Sequence 2 (Experimental): Paper migraine diary followed by AI-empowered voice-interactive chatbot
  Interventions: Device: Paper migraine diary; Device: AI-empowered voice-interactive chatbot

INTERVENTIONS:
Device: AI-empowered voice-interactive chatbot — Participants will interact with the chatbot on a daily basis to record their migraine experiences. They will be asked to initiate a conversation with the chatbot whenever they experience a migraine attack and provide the required information, including the date and time of the attack, presence of aura, migraine intensity, accompanying symptoms, triggers, and medication use. The chatbot will engage participants in a conversation to collect these data points and store them securely within the chatbot system.
  Arms: Sequence 1
Device: Paper migraine diary — Participants will manually document their migraine experiences on the paper migraine diary, including the date and time of the attack, presence of aura, migraine intensity, accompanying symptoms, triggers, and medication use.
  Arms: Sequence 1
Device: Paper migraine diary — Participants will manually document their migraine experiences on the paper migraine diary, including the date and time of the attack, presence of aura, migraine intensity, accompanying symptoms, triggers, and medication use.
  Arms: Sequence 2
Device: AI-empowered voice-interactive chatbot — Participants will interact with the chatbot on a daily basis to record their migraine experiences. They will be asked to initiate a conversation with the chatbot whenever they experience a migraine attack and provide the required information, including the date and time of the attack, presence of aura, migraine intensity, accompanying symptoms, triggers, and medication use. The chatbot will engage participants in a conversation to collect these data points and store them securely within the chatbot system.
  Arms: Sequence 2

SUMMARY:
The goal of this randomized crossover trial is to examine whether the AI-empowered chatbot will effectively collect comprehensive migraine feature data and demonstrate higher compliance, accuracy, utilization, acceptability, feasibility, and validity in migraine feature tracking compared to traditional paper-based migraine diaries among Hong Kong women with migraine.

Participants will use different tools (AI-empowered voice-interactive chatbot or paper migraine diary) for migraine tracking. Participants will be randomly allocated to one of two intervention sequences: (1) AI-empowered voice-interactive chatbot followed by paper migraine diary, or (2) paper migraine diary followed by AI-empowered voice-interactive chatbot. The study will consist of two intervention periods, each lasting one month, with a 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Meet diagnostic criteria for migraine according to ICHD-3
* Experiencing at least 2 headache days per month
* Living in Hong Kong
* Fluent in Cantonese
* Owning a smartphone with internet access
* Willing to provide informed consent

Exclusion Criteria:

* Individuals with severe cognitive impairments or communication difficulties
* Those unable to use a smartphone or the chatbot due to physical or mental limitations
* Using another alternative electronic migraine diary during recruitment or in the past 12 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
timeliness | At the end of each 1-month intervention period
  Timeliness will be defined as the proportion of migraine episodes recorded within 24 hours of onset. This measure will be derived from the data collected through the chatbot and paper diary.
Completeness | At the end of each 1-month intervention period
  Completeness will be defined as the proportion of diary entries with all required migraine-related information fully recorded. This measure will be derived from the data collected through the chatbot and paper diary.
Missed episodes | At the end of each 1-month intervention period
  Missed episodes will be defined as the proportion of migraine episodes not recorded; the number of missed episodes in each period will be obtained at the end-of-period questionnaire
Accuracy | At the end of each 1-month intervention period
  Accuracy will be defined as the proportion of diary entries in which all required migraine-related fields were recorded correctly. Accuracy will be adjudicated by assessing the consistency between migraine features recorded using the chatbot or paper diary and those reported during end-of-period online interviews with study staff. Discrepancies will be documented; records will be not altered for primary analyses. During these interviews, researchers will summarise the participant's recorded migraine information for that period, regardless of modality, and ask the participant to identify any errors.

SECONDARY OUTCOMES:
Utilization | At the end of each 1-month intervention period
  Utilization will be evaluated using the Chinese version of the System Usability Scale (SUS), a widely used and validated 10-item questionnaire that assesses the usability of a system on a 5-point Likert scale. The SUS yields a single score ranging from 0 to 100, with higher scores indicating better usability. Specifically, chatbot utilization will be objectively assessed using system-generated data, such as the number of logins, user-initiated conversations, and user responses.
Acceptability | At the end of each 1-month intervention period
  Acceptability will be measured using the validated Chinese version of Technology Acceptance Model (TAM) scale, an 11-item questionnaire on a 7-point Likert scale with higher scores indicating greater acceptance.
Usage | At the end of each 1-month intervention period
  Usage will be assessed by the number of uses (entries) per tool.
Time per recording | At the end of each 1-month intervention period
  Time required to record each migraine episode, using system-logged durations for the chatbot and self-recorded start and finish times for the paper diary.
Validity | At the end of each 1-month intervention period
  The validity of the migraine data collected through the chatbot and paper diary will be assessed using convergent validity and divergent validity. Convergent validity will be evaluated by examining the correlation between migraine frequency and severity recorded using the chatbot or paper diary and the Chinese version of the Migraine Disability Assessment (MIDAS) scores (0 to 270, higher scores indicating greater migraine-related disability). Divergent validity will be assessed by analyzing the correlation between migraine frequency and severity and the Chinese version of the Brief Self-Control Scale (7 to 35, with a higher score indicating greater self-control).

CONTACTS AND LOCATIONS:
Overall Officials: Yao Jie Xie, PhD, Principal Investigator — The Hong Kong Polytechnic Univeristy
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, HONG KONG, Hong Kong

IPD SHARING:
Plan to Share IPD: No